CLINICAL TRIAL: NCT03825978
Title: Evaluation of Efficacy of Counseling for Prenatal Screening and Diagnostic Tests on Pregnant Women's Decisional Conflict, Being Sure of the Decision, Anxiety Levels and Attitudes Towards the Tests: A Randomised Controlled Clinical Study
Brief Title: Efficacy of Counseling for Prenatal Screening and Diagnostic Tests on Pregnant Women: Randomised Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Ilknur Yesilcinar, PhD. RN., Principal Investigator, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Ilknur Yesilcinar
Record Dates: First submitted 2019-01-23; First posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Decision Making; Chromosome Abnormality; Anxiety; Knowledge, Attitudes, Practice
Keywords: prenatal genetic screening; prenatal diagnosis; counseling; decision; anxiety; nursing
MeSH Terms: conditions — Chromosome Aberrations; Anxiety Disorders; Behavior | interventions — Genetic Counseling; Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): An individual and comprehensive prenatal genetic counseling was given to all pregnant women in the intervention group, including all screening tests and diagnostic tests for prenatal diagnosis and screening tests at the first antenatal visit.
  Interventions: Behavioral: Prenatal Genetic Counseling
- Control (No Intervention): There was no intervention from the first antenatal visit in the control group. Routine clinical information was given about prenatal screening and diagnostic tests.

INTERVENTIONS:
Behavioral: Prenatal Genetic Counseling — In this study prenatal genetic screening counseling was provided from the begining of the pregnancy, different from the other studies in the literature. In the literature, most of the study evaluated pregnant women's anxiety, information status about the test and decisional conflicts, only prenatal screening process or prenatal diagnosis process. In this study pregnant women were evaluated both in prenatal screening test and prenatal diagnosis procedures.
  Other Names: Counseling
  Arms: Intervention

SUMMARY:
The aim of this study was to evaluate the effect of counseling for prenatal screening and diagnostic tests on pregnant women's decisional conflict, being sure of the decision, anxiety levels, and attitudes towards the tests. This prospective randomized controlled intervention study was conducted between the dates June 2017 and March 2018 in a training and research hospital, department of obstetrics and gynecology. The sample of the study consisted of 210 pregnant women who took antenatal care between the 8-11th gestational weeks of whom 112 were in the intervention group and 98 were in the control group. The data were collected by using Data Collection Form, The State-Trait Anxiety Inventory (STAI I-II), Decisional Conflict Scale (DCS), Sure Scale (SURE), Knowledge Evaluation Form about Prenatal Genetic Screening and Diagnostic Tests, Prenatal Counseling Satisfaction Form, Decision Satisfaction Form and Attitudes towards the tests Scale. The study carried out in two stages. In the first stage; women's data were collected before and after participating prenatal genetic screening tests. After the results of the screening test were taken, the data were collected again. Counseling was provided for 112 pregnant women about prenatal screening and diagnostic tests before participating tests. Routine clinical information was given for 98 pregnant women who were in control group. Both groups were pre and post-tested at the same times. In the second phase, pregnant women who had diagnostic tests were evaluated. Counseling for prenatal genetic diagnosis tests was provided for 31 pregnant women in inetervetion group women and routine clinical information was providen for 26 pregnant women who were in control group. Data were collected again with data collection tools before and after the diagnostic test.

DETAILED DESCRIPTION:
Pregnant Women Who Had Only Prenatal Genetic Screening Tests In intervention group, pregnant women, who were in 8-11th gestational weeks, before prenatal genetic counseling, answered the questions in "Descriptive Features Data Collection Form", "Decisional Conflict Scale", "The State-Trait Anxiety Inventory scale", "Information Evaluation Form about Prenatal Screening Tests ","Decision Satisfaction Scale", "Attitudes towards the tests Scale". Later, individual interviews were made with pregnant women education was given with slide show about prenatal diagnosis and screening tests to pregnant women. In addition a training brochure which was prepared by the researcher was given to the pregnant women. It took about 20 minutes for the data collection forms to be answered and counseling was took about 25 minutes. After counseling, pregnant women were interviewed again at 14th week. The pregnant women were asked whether they had a screening test and the results were recorded. Then pregnant women were answered "Decisional Conflict Scale", "The State-Trait Anxiety Inventory scale", "Information Evaluation Form about Prenatal Screening Tests ","Decision Satisfaction Scale", "Attitudes towards the tests Scale" again. At the following antenatal visits (16-20th weeks), the pregnant women were asked whether they had triple, quadruple or NIPT and the test results were recorded in the data collection form. At the end of the 20th week, the data collection process of pregnant women who did not have any problems related to fetus and who were recommended to continue routine follow-up was terminated. In control group pregnant women answered same data collection forms in same weeks, but counseling was not given to this group. For this group routine clinical procedure was performed.

Pregnant Women Who Had Also Prenatal Genetic Diagnostic Tests Prenatal genetic diagnostic tests were recommended to pregnant women who had high risk results according to prenatal screening test. Pregnant women with high risk and diagnostic test were referred to genetic consultation in both intervention and control groups. After genetic consultation, pregnant women were answered "Decisional Conflict Scale", "The State-Trait Anxiety Inventory scale", "Information Evaluation Form about Prenatal Diagnostic Tests", "Decision Satisfaction Scale", "Attitudes towards the tests Scale". Then specific counseling was given to invasive test recommended by the doctor. The pregnant woman was asked if she would like to have a diagnostic test and if she didn't want to, the reason was recorded in the data collection form.

If the pregnant woman decided to have a diagnostic test, "The State-Trait Anxiety Inventory scale" was applied again after the procedure. Then pregnant women were interviewed again after about three weeks and their results were evaluated and they answered "Decisional Conflict Scale", "Information Evaluation Form about Prenatal Diagnostic Tests", "Decision Satisfaction Scale", "Attitudes towards the tests Scale". Their decision about to continue or terminate pregnancy was recorded in the data collection form. In control group pregnant women answered same data collection forms in same weeks, but counseling was not given to this group. For this group routine clinical procedure was performed.

ELIGIBILITY:
Inclusion Criteria:

* taking first antenatal follow-up in 8-11. gestational weeks in where the study is conducted to have a single pregnancy
* to continue take the antenatal care in the hospital where the research was conducted
* at least primary school graduation,
* voluntary to participate the research.

Exclusion Criteria:

* want to exit from the study at her own request
* continue to antenatal follow-up in another hospital.

Ages: 19 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women was evaluated in this study
Enrollment: 260 (Actual)
Dates: Start 2017-06-10 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
Anxiety | In 8-11th gestational weeks
  The State Anxiety Scale evaluates the current state of anxiety. The expressions (1) in the articles are rated as (2) slightly, (3) very, (4) completely, and the scale is answered by marking the ones that meet the current situation of the person. The total point value obtained from scale may vary between 20 and 80 points. High score indicates high anxiety level and low score indicates low anxiety level
Decisional Conflict | In 8-11th gestational weeks
  Pregnant women's decisional conflict scale points: 5-point Likert type and 16 questions.
  Each item varies between "Strongly Agree ıy and" Strongly Disagree Her. Each item contains direct expressions, and I absolutely agree with = 0 points, Agree = 1 points, Undecided = 2 points, Disagree = 3 points and Strongly Disagree = 4 points. While calculating the total scale score; points are awarded to all items. The score is divided by the total number of items and is multiplied by 25 and the scale score is obtained. There is no cut-off point in the scale evaluating decision conflict scores. As the score obtained from the scale increases, the level of decision conflict increases.
SURE Scale | In 8-11th gestational weeks
  Pregnant women's SURE Scale points: It is double likert type. Items Yes = 1 point No = 0 points. Zero points mean that there is a very high decision-making conflict, while 4 points mean that there is no conflict. Scores of 3 points or less indicate a conflict of interest.
Knowledge Form About Prenatal Genetic Screening and Diagnostic Tests | In 8-11th gestational weeks
  Pregnant Women's Prenatal Genetic Screening and Diagnostic Tests Form points: The information evaluation form for prenatal screening tests was developed by the researcher as a result of literature review. The information evaluation form for prenatal screening tests consists of 12 statements. The aim of the prenatal screening tests is to provide information about the diseases, the weeks of screening tests, risk values and what they mean. For each phrase there are yes, I don't know and no options.Twelve is Highest, 0 is the lowest scores.
Attitudes Towards The Tests Scale | In 8-11th gestational weeks
  Pregnant women's Attitudes Towards The Tests scale points: Good idea to participate in testing for prenatal screening and diagnostic tests on the scale (7 points), bad idea (1 point); useful (7 points), not useful (1 point); harmful (1 point), not harmful (7 points); a bad idea (1 point), not a bad idea (7 points) were asked to rank between 1 and 7 points. One point represents negative attitude and 7 points represent a very positive attitude. According to the opinions of the pregnant women about the prenatal screening and diagnostic tests, it was stated that they could give the expressions between 1 and 7, and they were asked to answer the scale. The highest score to be obtained from this scale is 28 and the lowest score is 4.
Decision Satisfaction Form | In 8-11th gestational weeks
  Pregnant women's Decision Satisfaction Form points: Developed by researchers. The participants were asked to evaluate whether they were satisfied with their decisions, to make an informed decision, to make informed decisions, to make the same decision if they had experienced the same situation again. In this form, which consists of five questions and has a five-point Likert type, the expressions are evaluated with 5 (strongly agree), 4 (agree), 3 (unclear), 2 (disagree), 1 (strongly disagree) options. The highest 25 points are the lowest 5 points. High score shows high satisfaction.

SECONDARY OUTCOMES:
Anxiety | In 13-14th gestational weeks
  The State Anxiety Scale evaluates the current state of anxiety. The expressions (1) in the articles are rated as (2) slightly, (3) very, (4) completely, and the scale is answered by marking the ones that meet the current situation of the person. The total point value obtained from scale may vary between 20 and 80 points. High score indicates high anxiety level and low score indicates low anxiety level
Decisional Conflict Scale | In 13-14th gestational weeks
  Pregnant women's decisional conflict scale points: 5-point Likert type and 16 questions.
  Each item varies between "Strongly Agree ıy and" Strongly Disagree Her. Each item contains direct expressions, and I absolutely agree with = 0 points, Agree = 1 points, Undecided = 2 points, Disagree = 3 points and Strongly Disagree = 4 points. While calculating the total scale score; points are awarded to all items. The score is divided by the total number of items and is multiplied by 25 and the scale score is obtained. There is no cut-off point in the scale evaluating decision conflict scores. As the score obtained from the scale increases, the level of decision conflict increases.
SURE Scale | In 13-14th gestational weeks
  Pregnant women's SURE Scale points: It is double likert type. Items Yes = 1 point No = 0 points. Zero points mean that there is a very high decision-making conflict, while 4 points mean that there is no conflict. Scores of 3 points or less indicate a conflict of interest.
Knowledge Form About Prenatal Genetic Screening and Diagnostic Tests | In 13-14th gestational weeks
  Pregnant women's Knowledge About Prenatal Genetic Screening and Diagnostic Tests Form Points: The information evaluation form for prenatal screening tests was developed by the researcher as a result of literature review. The information evaluation form for prenatal screening tests consists of 12 statements. The aim of the prenatal screening tests is to provide information about the diseases, the weeks of screening tests, risk values and what they mean. For each phrase there are yes, I don't know and no options. Twelve is Highest, 0 is the lowest scores.
Attitudes Towards The Tests Scale | In 13-14th gestational weeks
  Pregnant women's Attitudes Towards The Tests Scale Points: Good idea to participate in testing for prenatal screening and diagnostic tests on the scale (7 points), bad idea (1 point); useful (7 points), not useful (1 point); harmful (1 point), not harmful (7 points); a bad idea (1 point), not a bad idea (7 points) were asked to rank between 1 and 7 points. One point represents negative attitude and 7 points represent a very positive attitude. According to the opinions of the pregnant women about the prenatal screening and diagnostic tests, it was stated that they could give the expressions between 1 and 7, and they were asked to answer the scale. The highest score to be obtained from this scale is 28 and the lowest score is 4.
Decision Satisfaction Form | In 13-14th gestational weeks
  Pregnant Women's Decision Satisfaction Form Points: Developed by researchers. The participants were asked to evaluate whether they were satisfied with their decisions, to make an informed decision, to make informed decisions, to make the same decision if they had experienced the same situation again. In this form, which consists of five questions and has a five-point Likert type, the expressions are evaluated with 5 (strongly agree), 4 (agree), 3 (unclear), 2 (disagree), 1 (strongly disagree) options. The highest 25 points are the lowest 5 points. High score shows high satisfaction.

OTHER OUTCOMES:
Decisional Conflict Scale | Before performing prenatal genetic diagnostic test at 16 weeks for who had amniosenthesis, 12 weeks for who had corionic villus sampling (For Women who had diagnostic tests)
  Pregnant women's Decisional Conflict Scale points: 5-point Likert type and 16 questions.
  Each item varies between "Strongly Agree ıy and" Strongly Disagree Her. Each item contains direct expressions, and I absolutely agree with = 0 points, Agree = 1 points, Undecided = 2 points, Disagree = 3 points and Strongly Disagree = 4 points. While calculating the total scale score; points are awarded to all items. The score is divided by the total number of items and is multiplied by 25 and the scale score is obtained. There is no cut-off point in the scale evaluating decision conflict scores. As the score obtained from the scale increases, the level of decision conflict increases.
SURE Scale | Before performing prenatal genetic diagnostic test at 16 weeks for who had amniosenthesis, 12 weeks for who had corionic villus sampling (For Women who had diagnostic tests)
  Pregnant women's SURE Scale points: It is double likert type. Items Yes = 1 point No = 0 points. Zero points mean that there is a very high decision-making conflict, while 4 points mean that there is no conflict. Scores of 3 points or less indicate a conflict of interest.
Knowledge Form About Prenatal Genetic Diagnostic Tests | Before performing prenatal genetic diagnostic test at 16 weeks for who had amniosenthesis, 12 weeks for who had corionic villus sampling (For Women who had diagnostic tests)
  Pregnant women's Knowledge About Prenatal Genetic Diagnostic Tests Form points: The information evaluation form for prenatal diagnostic tests was developed by the researcher as a result of literature review. The information evaluation form for prenatal diagnostic tests consists of 10 statements. The aim of this form is to provide information about the diseases, the weeks of diagnostic tests, tests' aims and what they mean. For each phrase there are yes, I don't know and no options. Ten is Highest, 0 is the lowest scores.
Attitudes Towards The Tests Scale | Before performing prenatal genetic diagnostic test at 16 weeks for who had amniosenthesis, 12 weeks for who had corionic villus sampling (For Women who had diagnostic tests)
  Pregnant women's Attitudes Towards The Tests Scale points: Good idea to participate in testing for prenatal screening and diagnostic tests on the scale (7 points), bad idea (1 point); useful (7 points), not useful (1 point); harmful (1 point), not harmful (7 points); a bad idea (1 point), not a bad idea (7 points) were asked to rank between 1 and 7 points. One point represents negative attitude and 7 points represent a very positive attitude. According to the opinions of the pregnant women about the prenatal screening and diagnostic tests, it was stated that they could give the expressions between 1 and 7, and they were asked to answer the scale. The highest score to be obtained from this scale is 28 and the lowest score is 4.
Decision Satisfaction Form | Before performing prenatal genetic diagnostic test at 16 weeks for who had amniosenthesis, 12 weeks for who had corionic villus sampling (For Women who had diagnostic tests)
  Pregnant women's Decision Satisfaction Form points:Developed by researchers. The participants were asked to evaluate whether they were satisfied with their decisions, to make an informed decision, to make informed decisions, to make the same decision if they had experienced the same situation again. In this form, which consists of five questions and has a five-point Likert type, the expressions are evaluated with 5 (strongly agree), 4 (agree), 3 (unclear), 2 (disagree), 1 (strongly disagree) options. The highest 25 points are the lowest 5 points. High score shows high satisfaction.
Anxiety | Before performing prenatal genetic diagnostic test at 16 weeks for who had amniosenthesis, 12 weeks for who had corionic villus sampling (For Women who had diagnostic tests)
  The State Anxiety Scale evaluates the current state of anxiety. The expressions (1) in the articles are rated as (2) slightly, (3) very, (4) completely, and the scale is answered by marking the ones that meet the current situation of the person. The total point value obtained from scale may vary between 20 and 80 points. High score indicates high anxiety level and low score indicates low anxiety level
Anxiety | After performing prenatal genetic diagnostic test at 20th weeks for who had amniosenthesis, 16 weeks for who had corionic villus sampling(For Women who had diagnostic tests)
  The State Anxiety Scale evaluates the current state of anxiety. The expressions (1) in the articles are rated as (2) slightly, (3) very, (4) completely, and the scale is answered by marking the ones that meet the current situation of the person. The total point value obtained from scale may vary between 20 and 80 points. High score indicates high anxiety level and low score indicates low anxiety level
Decisional Conflict Scale | After performing prenatal genetic diagnostic test at 20th weeks for who had amniosenthesis, 16 weeks for who had corionic villus sampling(For Women who had diagnostic tests)
  Pregnant women's Decisional Conflict Scale points: 5-point Likert type and 16 questions.
  Each item varies between "Strongly Agree ıy and" Strongly Disagree Her. Each item contains direct expressions, and I absolutely agree with = 0 points, Agree = 1 points, Undecided = 2 points, Disagree = 3 points and Strongly Disagree = 4 points. While calculating the total scale score; points are awarded to all items. The score is divided by the total number of items and is multiplied by 25 and the scale score is obtained. There is no cut-off point in the scale evaluating decision conflict scores. As the score obtained from the scale increases, the level of decision conflict increases.
SURE Scale | After performing prenatal genetic diagnostic test at 20th weeks for who had amniosenthesis, 16 weeks for who had corionic villus sampling(For Women who had diagnostic tests)
  Pregnant women's SURE Scale points: It is double likert type. Items Yes = 1 point No = 0 points. Zero points mean that there is a very high decision-making conflict, while 4 points mean that there is no conflict. Scores of 3 points or less indicate a conflict of interest.
Knowledge Form About Prenatal Genetic Diagnostic Tests | After performing prenatal genetic diagnostic test at 20th weeks for who had amniosenthesis, 16 weeks for who had corionic villus sampling(For Women who had diagnostic tests)
  Pregnant women's Knowledge About Prenatal Genetic Diagnostic Tests Form points: The information evaluation form for prenatal diagnostic tests was developed by the researcher as a result of literature review. The information evaluation form for prenatal diagnostic tests consists of 10 statements. The aim of this form is to provide information about the diseases, the weeks of diagnostic tests, tests' aims and what they mean. For each phrase there are yes, I don't know and no options. Ten is Highest, 0 is the lowest scores.
Attitudes Towards The Tests Scale | After performing prenatal genetic diagnostic test at 20th weeks for who had amniosenthesis, 16 weeks for who had corionic villus sampling(For Women who had diagnostic tests)
  Pregnant women's Attitudes Towards The Tests Scale points: Good idea to participate in testing for prenatal screening and diagnostic tests on the scale (7 points), bad idea (1 point); useful (7 points), not useful (1 point); harmful (1 point), not harmful (7 points); a bad idea (1 point), not a bad idea (7 points) were asked to rank between 1 and 7 points. One point represents negative attitude and 7 points represent a very positive attitude. According to the opinions of the pregnant women about the prenatal screening and diagnostic tests, it was stated that they could give the expressions between 1 and 7, and they were asked to answer the scale. The highest score to be obtained from this scale is 28 and the lowest score is 4.
Decision Satisfaction Form | After performing prenatal genetic diagnostic test at 20th weeks for who had amniosenthesis, 16 weeks for who had corionic villus sampling(For Women who had diagnostic tests)
  Pregnant women's Decision Satisfaction Form points: Developed by researchers. The participants were asked to evaluate whether they were satisfied with their decisions, to make an informed decision, to make informed decisions, to make the same decision if they had experienced the same situation again. In this form, which consists of five questions and has a five-point Likert type, the expressions are evaluated with 5 (strongly agree), 4 (agree), 3 (unclear), 2 (disagree), 1 (strongly disagree) options. The highest 25 points are the lowest 5 points. High score shows high satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: İlknur Yeşilçınar, PhD. RN., Study Director — Health Science University; Gülten Güvenç, Assoc. Prof., Study Director — Health Science University
Locations (2):
- Turkey (Türkiye) (2):
  - Health Science University, Ankara
  - University Of Health Sciences, Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin L, Gitsels-van der Wal JT, de Boer MA, Vanstone M, Henneman L. Introduction of non-invasive prenatal testing as a first-tier aneuploidy screening test: A survey among Dutch midwives about their role as counsellors. Midwifery. 2018 Jan;56:1-8. doi: 10.1016/j.midw.2017.09.008. Epub 2017 Sep 24. PMID 29024868
- [Background] Amel S.H., Ali A, Hassan S.A, Momtaz M., Abdelhaleem Z., Negm S. Impact of A Structured Prenatal Counseling on Anxiety Level Among Women Undergoing Amniocentesis. American Journal of Research Communication, 2014; 2(6): 97-108} www.usa-journals.com, ISSN: 2325-4076.
- [Result] Long S, O'Leary P, Lobo R, Dickinson JE. Women's Understanding and Attitudes towards Down Syndrome and Other Genetic Conditions in the Context of Prenatal Screening. J Genet Couns. 2018 Jun;27(3):647-655. doi: 10.1007/s10897-017-0167-7. Epub 2017 Oct 24. PMID 29067542